CLINICAL TRIAL: NCT05011656
Title: Blood Purification for the Treatment of Critically Ill Patients With Pathogen Associated Shock: A Multicenter, Randomized Controlled Feasibility Trial
Brief Title: Blood Purification for the Treatment of Pathogen Associated Shock
Acronym: PURIFY-RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ExThera Medical Corporation (Industry)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PURIFY Multi-center RCT
Record Dates: First submitted 2021-07-29; First posted 2021-08-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Septic Shock
Keywords: pathogen associated shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either Arm 1: Seraph 100 treatment plus 'State of the Art' or Arm 2: 'State of the Art' care alone. "State of the Art care" will be defined as the treatment algorithms outlined in the Surviving Sepsis Campaign for the treatment of septic shock, available at https://www.sccm.org/SurvivingSepsisCampaign/Home
Masking Description: Unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 1- Seraph-100 plus State of the Art Care (Experimental): The Seraph 100 Filter is a single use, disposable column packed with ultra-high molecular weight polyethylene beads which have been modified to contain endpoint attached heparin on the surface. Seraph 100 is an extracorporeal broad-spectrum sorbent hemoperfusion device for reduction of pathogens from the bloodstream. It is intended for use with standard, commercially available bloodlines compatible with the pump system used. Female Luer connectors are required to connect to the Seraph 100 blood ports.
  Interventions: Device: Seraph-100 + State of the Art Care
- 2 - State of the Art Care (Active Comparator): "State of the Art care"is defined as the treatment algorithms outlined in the Surviving Sepsis Campaign for the treatment of septic shock, available at https://www.sccm.org/SurvivingSepsisCampaign/Home
  Interventions: Device: State of the Art Care

INTERVENTIONS:
Device: Seraph-100 + State of the Art Care — Seraph® 100 Microbind® Affinity Blood Filter (Seraph 100) manufactured by ExThera Medical Corporation in Martinez, CA. The Seraph 100 filter has been designed and manufactured to reduce residual risks as much as possible to ensure safe usage. Literature search results concluded that heparin-coated medical devices are safe and decrease platelet adhesion without affecting the adsorption of major adhesive proteins. The efficacy, safety, and risk-benefit data of the studies suggest that Seraph 100 is also safe and potentially beneficial by reducing the rate of thrombosis, without its use entailing a risk for patients. The achieved results from the above-mentioned testing and studies support the performance and safety of Seraph 100 consistent with the intended use. ExThera Medical concludes that the known and potential benefits of Seraph 100, when used to treat patients with pathogen associated shock, outweigh the known and potential risks when used according to the intended use.
  Arms: 1- Seraph-100 plus State of the Art Care
Device: State of the Art Care — "State of the Art care"is defined as the treatment algorithms outlined in the Surviving Sepsis Campaign for the treatment of septic shock, available at https://www.sccm.org/SurvivingSepsisCampaign/Home
  Arms: 2 - State of the Art Care

SUMMARY:
This study is a multi-center, randomized controlled feasibility trial to evaluate the initial safety and efficacy of a novel extracorporeal blood purification (EBP) therapy in critically ill patients with pathogen associated shock across 15 U.S. sites. Adults (18 years old and older) admitted to the ICU with all of the following:

• Pathogen associated shock defined as:

* The need for vasopressors to maintain mean arterial pressure (MAP) ≥ 65 mmHg despite adequate fluid resuscitation
* Presence of a pathogen detected in the bloodstream within 72 hours of screening using commercially available in-vitro diagnostic testing

DETAILED DESCRIPTION:
Patients meeting the eligibility criteria will be randomized to receive either treatment with the investigational device (Seraph 100) + 'State of the Art' care versus 'State of the Art' care alone. This study is a multi-center, un-blinded, randomized controlled feasibility trial to evaluate the initial safety and efficacy of Seraph 100 in critically ill patients with pathogen associated shock across 15 US sites. This study will not be done in a blinded fashion from either the patient or caregiver perspective given: 1) the need for invasive, central line placement, and 2) to ensure that limited hospital resources (e.g., hemodialysis machines) are available for patients that require therapy. While the study trial will not be conducted in a blinded fashion, the members of the study team that do the data analysis will be blinded.

The target population is adults (18 years old and older) admitted to the ICU with all of the following:

* Pathogen associated shock AND
* The need for vasopressors at any dose to maintain mean arterial pressure (MAP) ≥ 65 mm Hg despite adequate fluid resuscitation.

Study Arms: Patients will be randomized to receive either Arm 1: Seraph 100 treatment plus 'State of the Art' or Arm 2: 'State of the Art' care alone. "State of the Art care" will be defined as the treatment algorithms outlined in the Surviving Sepsis Campaign for the treatment of septic shock, available at https://www.sccm.org/SurvivingSepsisCampaign/Home.

Study Randomization and stratification: Patients who qualify will be immediately randomized. The study will randomize patients 2:1 to investigational product plus 'State of the Art' care and 'State of the Art' alone, respectively. Upon randomization, patients will be stratified by age (≥65 and <65). While ideally, the research team would stratify by other variables (to include demographics, causative pathogen, GCS, SOFA, associated organ failure, and pre-existing conditions), given the small number of patients in this trial (particularly in the control group) this is not possible.

The Seraph 100 Microbind® Affinity Blood Filter (Seraph 100) manufactured by ExThera Medical Corporation in Martinez, CA.

Investigational Treatment Duration for Seraph 100: A sufficient blood flow rate and exposure of the patient's blood to the Seraph 100 adsorption media will optimize the treatment success with a target total filtered blood volume of 100L per day. Based on the target total filtered blood volume of 100L, the average treatment duration and blood flow rates are captured below:

Average Blood Flow Rate Treatment Duration 350 ml/min 5 hours 300 ml/min 6 hours 250 ml/min 7 hours 200 ml/min 8 hours

* At an average blood flow of 350mL/min, this would translate to almost 5 hours of treatment time; an average of 200mL/min would mean a treatment time of 8 hours.
* Treatments will occur daily for up to 4 consecutive days or until all of the following criteria are met:

  * Vasopressor-free for >24h
  * MAP≥65
* Treatments will be held if subjects are unable to tolerate extra-corporeal therapy (defined as MAP<65 despite fluids and vasopressors)

Patients will be assessed daily while hospitalized as part of routine, standard of care in the ICU. All patients enrolled in this study will undergo clinical efficacy, safety, and laboratory assessments. Blood, urine, and respiratory samples will be obtained at baseline, Day 1 (pre/post treatment) through Day 4, Day 7, and Day 28. Demographic and baseline clinical parameters will be recorded at the time of randomization. Pertinent clinical parameters will be recorded hourly for the first 96 hours, once on day 7, and once on day 28. SOFA scores will be recorded daily for the first 7 days. Outcomes data will be recorded on day 28 and at the time of hospital discharge or death. Patient status will be assessed at 30, 60, and 90 days to include vital signs, physical examination, adverse event evaluation, and a targeted medication review. Survival status will be assessed 90 days after enrollment (if the patient is no longer hospitalized).

The first 10 patients randomized to interventional therapy, as well as the first 5 patients randomized to the control group, will undergo additional pharmacokinetic (PK) evaluation of antimicrobial removal by the filter treatment. These first 15 total patients enrolled must also meet all requirements for the main portion of the study.

As part of the initial PK study, the Data Safety Monitoring Board (DSMB) will also review safety data after the first 5 device patients consented and treated. Safety and PK data will also be reviewed after the first 10 device patients are consented and treated. If there are significant safety concerns after DSMB review, the sponsor will immediately pause the trial and communicate the information with the FDA.

The PK results of the first 10 treatment patients will be reported to FDA for review to confirm the proposed dosing prior to commencing enrollment of the remaining subjects for a total of 60 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to an ICU with pathogen associated shock defined as:

   * The need for vasopressors to maintain mean arterial pressure (MAP) ≥ 65 mmHg despite adequate fluid resuscitation, AND
   * Presence of a pathogen detected in the bloodstream within 72 hours of screening using commercially available in-vitro diagnostic testing
2. Male or non-pregnant female adult
3. At least 18 years of age at time of enrollment

Exclusion Criteria:

1. Pregnant or breast feeding
2. Anticipated transfer to another hospital (that is not a study site) within 72 hours for any reason
3. Not anticipated to survive more than 24 hours
4. Known allergy to heparin sodium
5. Patients who cannot tolerate placement of double-lumen catheter
6. High risk of bleeding (platelet count <50mm3 or International Normalized Ratio (INR) >2) unless adequate line for treatment already placed (e.g. ECMO or RRT/CRRT)
7. Inability to tolerate extracorporeal therapy (defined as MAP<65 despite fluids and vasopressors)
8. Advanced cancer (defined as stage IV) with life expectancy of less than 30 days
9. Unable to obtain informed consent from either patient or legally authorized representative (LAR)
10. Hypotension and volume depletion due to etiologies other than sepsis.
11. Neutropenia with an absolute neutrophil count <500mm3
12. Patients must be treated with one of the antimicrobial agents listed in the Antimicrobial Management Guideline (Table 19). Patients who require treatment with an antimicrobial outside of this list while still receiving treatment with the investigational device must be excluded from the study.
13. If a patient enters the study and later requires a change in the antimicrobial agent used to one which is not listed in the Antimicrobial Management Guideline while still receiving treatment with the investigational device, that patient must be removed from this trial. Clinical data for any patient removed from the trial for this reason will continue to be collected for safety evaluation".
14. Patient is a prisoner or member of a different vulnerable population that should not be included in the study per the investigator or IRB/ethics committee.
15. Advanced directive for "Do Not Resuscitate".

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy - ICU-free days in the first 28 days | First 28 days
  Alive and not in the ICU (for at least a fulle 24 hours) in the first 28 days from the time of randomization
Safety - Adverse Events | Discharge from hospital
  SAEs and >/= grade 3 AEs per CTCAE v5 evaluated from enrollment until the end of hospitalization

SECONDARY OUTCOMES:
Mortality | 28 days
  Evaluate in-hospital mortality and mortality at 28 days
Ventilator-free days in the first 28 days | First 28 days
  Alive and free of mechanical ventilation (for at least a full 24 hours) in the first 28 days from the time of randomization
Vasopressor-free days in the first 28 days | First 28 days
  Alive and vasopressor-free for at least a 24-hour period in the first 28 days from the time of randomization
Kidney replacement therapy-free days in the first 28 days | First 28 days
  Alive and not on kidney replacement therapy for at least 72 hours.
Hospital Stay | through study completion, an average of 90 days
  number of days that the subject is hospitalized
Survival | through study completion, an average of 90 days
  Alive or dead 90 days after enrollment (if discharged from the hospital prior to 90 days after enrollment)

CONTACTS AND LOCATIONS:
Overall Officials: Lakhmir Chawla, MD, Study Chair — ExThera Medical
Locations (9):
- United States (9):
  - George Washington University, Washington D.C., District of Columbia
  - Southeast Georgia Health System, Inc., Brunswick, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Good Samaritan Hospital, Corvallis, Oregon
  - Trinity Health Mid Atlantic-SMMC, Langhorne, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Methodist Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio (UT Health San Antonio), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Following completion of the study, results of this research will be in a scientific journal. Data will be available immediately following publication, with no end date, with data sharing at the discretion of the sponsor.